CLINICAL TRIAL: NCT01370460
Title: Topical Tranexamic Acid and Acute Blood Loss in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 6669
Record Dates: First submitted 2011-06-03; First posted 2011-06-10 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Acute Blood Loss Anemia; Osteoarthritis, Knee
Keywords: Tranexamic Acid; Blood transfusion; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Experimental): Topical tranexamic acid (2g/100mL) applied during unilateral total knee arthroplasty.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): 100mL 0.9% NS, applied topically
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Topical tranexamic acid (2g/100mL 0.9% saline)
  Other Names: Cyklokapron
  Arms: Tranexamic Acid
Drug: Placebo — 100mL 0.9% sterile saline
  Arms: Placebo

SUMMARY:
This study aims to assess postoperative blood loss and transfusion rates in total knee replacement after one-time administration of topical tranexamic acid.

DETAILED DESCRIPTION:
Autologous (donor) blood transfusion is an expensive and common occurrence after total knee replacement. Published data puts this rate between 9 and 40% after primary unilateral total knee arthroplasty. There have been many proposed adjunctive measures to decrease intraoperative and postoperative blood loss during such surgery. Most of these include thrombin inhibition, so-called "minimally- invasive" techniques or instrumentation, or other adjunctive drugs. Hitherto, tranexamic acid, a specific drug that promotes part of the clotting cascade, has been used extensively in multiple areas of surgery with multiple studies evaluating its efficacy in cardiac surgery, spinal procedures, and as a dental swishing solution after tooth extraction. There have been small studies evaluating intravenous tranexamic acid and its effect on total knee replacement, with some promising results. The topical form of TA has been evaluated in only one prospective, randomized clinical trial with a significant decrease in postoperative blood loss and a trend towards decreased autologous blood transfusion rates. This study proposes to further evaluate tranexamic acid as an inexpensive and viable option for use in total knee arthroplasty. The topical form of the drug has been shown to achieve these hemostatic effects without increasing the risk of blood clots after surgery. Furthermore, the one aforementioned randomized clinical trial used a variety of postoperative deep vein thrombosis prophylaxis after surgery and introduced a potential confounding variable. A rigorous analysis of the effects of tranexamic acid demand a more standardized approach. Such a regimen is practiced at Henry Ford Hospital as all patients on the Adult Reconstruction service are placed on an identical dose of enoxaparin (a subcutaneous blood thinner) postoperatively for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over age eighteen
* Primary unilateral total knee arthroplasty at Henry Ford Hospital (Detroit, Michigan, United States) and Henry Ford West Bloomfield Hospital (West Bloomfield, Michigan, United States)

Exclusion Criteria:

* patient history of venous thromboembolic disease or coagulopathy
* use of anticoagulant medications within 7 days of surgery
* history of arterial embolic disease
* history of Class III or IV heart failure
* renal failure
* intraoperative cardiovascular, pulmonary, orthopaedic, or anesthetic complication (MI, intraoperative fracture, vasopressor support, emergent intubation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Laker, M.D., Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Good L, Peterson E, Lisander B. Tranexamic acid decreases external blood loss but not hidden blood loss in total knee replacement. Br J Anaesth. 2003 May;90(5):596-9. doi: 10.1093/bja/aeg111. PMID 12697586

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We planned on 50 patients in one treatment arm and 51 in another, resulting in 101 overall patients.
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 50 | 51
Completed | 50 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 51
  >=65 years | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 64.5 (8.2) | 65.75 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 39 | 70
  Male | 19 | 12 | 31
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss
Description: Preoperative and lowest postoperative hemoglobin. Blood loss was calculated taking change in hemoglobin as described (units g/dL) and converting to blood loss (mL) according to the formulas included in the papers cited in this entry (Good 2003 Br J Anesthesia; Nadler 1962 Surgery, http://www.ncbi.nlm.nih.gov/pubmed/21936146).
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 51 | 50
mL | 1293.1 (532.7) | 940.2 (327.1)

2. Secondary Outcome: Postoperative Transfusion Rate
Description: Number of patients with symptomatic (tachycardia, hypotension, presyncope) anemia of < 8.0g/dL hemoglobin, or any hemoglobin <7.0 g/dL, precipitated transfusion.
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 3 days
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 50 | 51
participants | 0 | 4

ADVERSE EVENTS:
Groups:
- Adverse Events Not Collected: Adverse Events Not Collected
Arm/Group | Adverse Events Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No